CLINICAL TRIAL: NCT05104658
Title: Heart Rehabilitation for All: A Feasibility Randomised Trial
Brief Title: Heart Rehabilitation for All
Acronym: HeRTA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Clinical Research and Prevention (Network)
Collaborators: Danish Heart Foundation (Other); Hvidovre University Hospital (Other); Albertslund Municipality (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-R136-A9125-22129
Record Dates: First submitted 2021-09-27; First posted 2021-11-03 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Ischemic Heart Disease; Cardiac Valve Surgery; Persistent Atrial Fibrillation; Heart Failure
Keywords: Heart disease; Heart rehabilitation
MeSH Terms: conditions — Myocardial Ischemia; Atrial Fibrillation; Heart Failure; Heart Diseases

STUDY DESIGN:
Intervention Model Description: The participants will be block randomised according to vulnerability to either the intervention or the control study arm
Masking Description: Masking is not possible as the primary outcome is participation in rehabilitation activities. However, health professionals at the hospital are allocated to either intervention or control group, to minimise cross-contamination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Usual rehabilitation: training (1 hour 2 times a week for 6 weeks), dietary training (2x3 hours), cardiac education (2x3 hours), referred to municipal rehabilitation: training (1 hour 2 times a week for 6-12 weeks), patient education (3x2 hours by a cardiac nurse and 1x2 hours by a dietician).
  In addition:
  * Information book on rehabilitation and physical activities in local community
  * 1:1 conversation with patient supporters from the Heart Association
  * Employer material on post-treatment and potential work adjustments
  * Support café for relatives
  * Supported transition to local sports associations
  * Motivating phone calls from physiotherapists supporting physical activities.
  In addition for patients with vulnerabilities:
  * patient education in small groups
  * pro-active counselling with a cardiac nurse, a psychologist, or a social worker from the Heart Association
  * paid transportation to the municipal rehabilitation Center
  Interventions: Other: Patient-targeted rehabilitation offers
- Control arm (No Intervention): Usual rehabilitation: training (1 hour 2 times a week for 6 weeks), dietary training (2x3 hours), cardiac education (2x3 hours), referred to municipal rehabilitation: training (1 hour 2 times a week for 6-12 weeks), patient education (3x2 hours by a cardiac nurse and 1x2 hours by a dietician).

INTERVENTIONS:
Other: Patient-targeted rehabilitation offers — In addition to usual rehabilitation services, patients in the intervention arm will receive patient-targeted rehabilitation offers to support the patients' participation and completion of their heart rehabilitation course.
  Arms: Intervention arm

SUMMARY:
Today, 50 % of cardiac patients do not participate in cardiac rehabilitation due difficulties in navigating and accessing rehabilitation activities.

HeRTA is a partnership project involving Center for Clinical Research and Prevention (CCRP), Hvidovre Hospital, Rehabilitation Center Albertslund and Copenhagen (municipalities), the Danish Heart Association, and local sports associations. A patient advisory board participate throughout the project to ensure a continued focus on patient interests.

The overall aim of HeRTA is to develop and test the feasibility of a new, sustainable model for rehabilitation supporting patients to take part in rehabilitation and promoting life-long activity for all patients with heart disease. To ensure equal access to rehabilitation some activities are open to all patients, while others are tailored specifically to patients with vulnerability.

The project unfolds in three phases: Development (1. January 1. 2020 - 14. November 2021): Partners and patients co-create content and procedures; Feasibility (15. November 2021 - 31. July 2023): The feasibility of the model is tested, and promising components are identified; Long-term follow-up and implementation (1. August 2023 - 31. December 2025): Long term effects are investigated and promising components are tested in new settings.

During the feasibility phase the investigators will examine whether the intervention activities are feasible, acceptable, and may have positive effects for patients with heart disease. The investigators use qualitative data on implementation and acceptability of intervention among partners and patients. An randomisered controlled trial (RCT) component will assess effects on patient participation rates, health, physical activity level, and life quality. Data is collected from practitioners and patients through focus groups, observations, field notes, questionnaires, and interviews.

Results will point to:

* innovative ways to organize integrated rehabilitation pathways.
* approaches to ensuring rehabilitation targeted at patient needs.

DETAILED DESCRIPTION:
1. Introduction

HeRTA is a partnership project conducted in close collaboration between hospital, municipality, patient organisation and local sports associations. A patient advisory board is involved throughout the project to ensure patient involvement including that decisions continuously focus on patient needs.

The overall aim of HeRTA is to develop and test the feasibility of a new, sustainable model for rehabilitation supporting vulnerable patients to take part in rehabilitation and promoting life-long activity for all patients with heart disease.

More specifically our goal is to:

* test if combined activities across sectors can increase the proportion of cardiac patients' participating in rehabilitation
* test if the model improves the maintenance of lifestyle changes and enhances physical and mental functioning, quality of life, and self-care capacity among cardiac patients

The project is organized in three phases:

1. An ongoing development phase, where all partners including the patient advisory board participate in a partnership and co-creation process to develop model content and collaboration procedures
2. A feasibility phase with a small scale RCT-component, where the investigators examine whether the intervention activities are feasible, acceptable, and may have positive effects for patients with heart disease
3. A long-term follow-up and implementation phase, in which sustainability of the intervention on patient activity is assessed and promising components are further tested.

2. Background Half a million Danes suffer from heart diseases. According to national guidelines rehabilitation should be offered to minimize consequences and prevent new cardiac episodes. Solid evidence exists on the benefits of multifaceted cardiac rehabilitation on patients' cardiovascular function, functional level, and survival.

Today, half of cardiac patients do not participate in rehabilitation. Structural barriers during the transition between hospital and municipality make it difficult to navigate rehabilitation activities. Additionally, the probability of being offered rehabilitation is lower if patients live alone, are unemployed, have a short education, a low income or suffer from several chronic conditions. Other barriers to participation are a poor financial situation, weak social relationships, logistic challenges, language difficulties, and cultural considerations. Even after having participated in rehabilitation programs, many patients struggle to maintain new lifestyle habits.

Despite health professionals' intentions to address vulnerability, vulnerable patients are overrepresented among those who do not receive a referral to rehabilitation, who do not participate in rehabilitation, and who do not complete rehabilitation activities.

3. Feasibility phase

During the development phase, partners and a patient advisory board has developed a model of combined activities aimed at creating a coherent rehabilitation course addressing needs among all patients with a special focus on patients with vulnerability.

Design, materials, and methods The investigators use qualitative data on implementation and acceptability of intervention among partners and patients. An RCT component will assess potential effects on patient participation rates, health, and life quality. The process evaluation will be guided by Normalization Process Theory and the Consolidated Framework for Implementation Research (CFIR). To ensure successful implementation and sustainability, partners will meet quarterly to evaluate experiences. In the initial three months, meetings are more frequent to allow for relevant adjustments. In the remaining inclusion period, strong rationale for changes should be provided to protect the potential of the study's RCT component. All changes in activities or procedures throughout the feasibility phase - including the rationale for adjustments - will be registered in field notes.

Registration of participation and sustainability Partners register patients' participation in all activities to monitor participation rates across sectors. Data from self-reported patient questionnaires are collected at baseline (background, and outcomes) and 3, and 6 months (outcomes, and participation in rehabilitation activities). At 12 and 24 months physical activity is assessed.

Qualitative data on patient experiences The research team conducts qualitative semi-structured interviews with 15-20 patients to uncover their experience of the overall process, contact with health care professionals, the match between activities and rehabilitation needs, patient involvement, and intersectoral coordination. Patients will be selected based on criteria for maximum variation. Both patients with high and low levels of participation will be selected for interviews.

Qualitative data on implementation among professionals Organizational characteristics and individual approaches among professionals will shape the implementation of activities. Field notes on adjustments in the intervention content, procedures, and changes in the context (e.g. organizational changes, changes in management/employees) will provide knowledge on the setting and the processes affecting the potential for the effect of the rehabilitation model. Observations and/or recordings of rehabilitation activities in hospital, municipality and Danish Heart Association will provide insight into the actual content of the activities and the fidelity of the implementation. Focus groups with involved partners will uncover the professional's experiences and reflections on screening and referral procedures, information exchange, intersectoral collaboration, and rehabilitation activities.

4. Evaluation

Descriptive analyses of the effect sizes The investigators will perform descriptive analyses of baseline characteristics. The primary outcome will be a) analyzed according to the intention-to-treat principle, b) sensitivity analyses of changes within/between the intervention and control groups will be carried out. If the power of data allows - explorative subgroup analyses will be carried out on those screened to be vulnerable. Estimated effect sizes will be calculated to inform future assessment of sample sizes in RCTs.

Qualitative evaluations All data from workshops, interviews, and focus groups will be audio-recorded and transcribed verbatim. Interview transcriptions and field notes will be analyzed using systematic text condensation described by Malterud. The analytical process will be inspired by principles from Collaborative Data Analysis.

Patients' experiences from the intervention The analysis will assess whether patients experience their treatment and rehabilitation course as an integrated and coordinated effort helping them to live with their heart disease. The analysis will nuance the quantitative analysis and assess whether the model succeeds in tailoring rehabilitation activities to individual needs. The full rehabilitation package is not necessary or relevant for all patients with heart disease. Patients with vulnerabilities may need elaborate support, while patients with resources may need less assistance. Rather they may need to be supported in using their local area and network to return to everyday life. In this analysis, gaps in the match between activities and patient needs will also be identified.

The implementation processes The analyses of organizational experiences will focus on the fit between the varying partnering institutions and the developed rehabilitation activities and collaboration procedures. Reach and fidelity of implementation will be assessed to provide relevant knowledge for interpreting and drawing conclusions on the potential of each intervention component.

Cost-effectiveness analyses A simple cost-effectiveness analyses will be carried out. This will be done by calculating a ratio where the denominator is the health gains measured by quality adjusted years of life (SF-12/SF-6D) and the numerator is the cost associated with the health gain obtained from the intervention, which will be the total cost of the intervention including resources used by the patients.

5. Project organization - A partnership

HeRTA is anchored in the Intersectoral Prevention Laboratory (IPL) with expertise in supporting intersectoral partnerships and intervention development and execution.

HeRTA is a partnership between researchers at CCRP, the IPL, the cardiac outpatient clinic at Hvidovre Hospital, Rehabilitation Center Albertslund and Copenhagen, and the Danish Heart Association. Local sports associations are part of the project at a collaborative level. The project receives sparring from an expert group and a patient advisory board.

Researchers at CCRP are Michaela Louise Schiøtz, Head of Section for Intersectoral Health Services Research; Hanne Birke, Ph.D., Postdoc with expertise in chronic disease (project manager); Karin Burns, a clinical coordinator with experience in supporting research in practice; Ida Foxvig, a research assistant with experience in partnerships and co-creation; Louise Meinertz Jakobsen, Ph.D., with expertise in interventions and rehabilitation.

An expert group provides professional feedback to the choice of research methods, outcome measurements, data collection, and analyses. Members are experts from Steno Diabetes Center Copenhagen, Hvidovre Hospital, Rigshospitalet, and the Immigrant Medical Clinic.

6. Ethics approval A data handling plan has been accepted by the Knowledge Center for Data Reviews, the Capital Region of Denmark (journal-nr.: P-2020-905). The National Committee of Health Research Ethics has approved the project (FSP 20035947).

7. Deliverables from the HeRTA feasibility study

The following deliverables are tangible outcomes of the project:

* Collaboration model across hospital, municipality, patient organization and local sports associations
* Feasible patient-targeted rehabilitation activities across sectors
* Identification of promising components to increase participation in rehabilitation and physical activity in local sports associations
* Tools to engage patients with vulnerability in rehabilitation

Communication plan The investigators provide an evidence-based contribution to the debate on cardiac rehabilitation and social inequalities in health and healthcare. The target groups for our communication are the research community; health professionals across sectors including leaders and key persons; civil society (e.g. patient organizations); and cardiac patients.

Findings will be presented in meetings, conferences, and written material, such as fact sheets and articles in peer-reviewed scientific journals and popular science journals and channels. The investigators will communicate through the Heart Foundation (Magazine and conference(s)) targeting cardiac patients and health professionals.

Perspectives Results from HeRTA will point to a model that is feasible and sustainable within the Danish healthcare system and forms a coherent rehabilitation pathway for people with cardiac disease. The model can be adjusted locally to fit the context in other rehabilitation locations and to ensure local stakeholder engagement. Our preliminary economic evaluation of financial cost and use of resources will operationalize the sustainability of the model.

HeRTA can form the basis for further targeted rehabilitation studies: a) rigorous RCT studies dissecting the effect of specific elements of the intervention that shows the greatest potential for positive benefits, and b) studies that test the generalizability across contexts to ensure transferability of results.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with ischaemic heart disease, cardiac valve surgery, persistent atrial fibrillation, or heart failure
2. Resident in Hvidovre Hospitals uptake area
3. Cognitively functional
4. Physically able to participate in rehabilitation activities

Exclusion Criteria:

* Patients, who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Participation in rehabilitation | Up to 20 months and two weeks
  The study's primary outcome is participation defined in three graduated participation levels:
  1. attending ≥ one activity (proactive counseling, patient education, smoking cessation, dietary counseling, physical exercise, local sports association activity).
  2. attending ≥ two activities (proactive counseling, patient education, smoking cessation, dietary counseling, physical exercise, local sports association activity).
  3. attending ≥ two activities (proactive counseling, patient education, smoking cessation, dietary counseling, physical exercise, local sports association activity) and reaching at least 50% turn up

SECONDARY OUTCOMES:
Sustained physical activity in leisure time | Up to 44 months + two weeks
  Data collected by questionnaires at baseline,3,6,12, and 24 months:
  Nordic Physical Activity Questionnaire-short (NPAQ): physical activities in leisure time.
Health-related quality of life | Up to 44 months + two weeks
  Data collected by questionnaire at baseline,3,6,12, and 24 months:
  The 12-Item Short Form Health Survey (SF-12):Physical and mental health summaries (PCS and MCS).
  1. General rating of health, score 1(best) to 5(worst)
  2. Limitation in moderate activities due to health, score 1(worst) to 3(best)
  3. Limited in climbing stairs due to health, score 1(worst) to 3(best)
  4. Accomplished less due to physical health, score 1(worst) to 5(best)
  5. Limited in daily activities due to physical health, score 1(worst) to 5(best)
  6. Accomplished less due to emotional problems, score 1(worst) to 5(best)
  7. Less careful due to emotional problems, score 1(worst) to 5(best)
  8. Pain affected normal work, score 1(best) to 5(worst)
  9. Felt calm and peaceful, score 1(best) to 5(worst)
  10. Had a lot of energy, score 1(best) to 5(worst)
  11. Felt down and depressed,score 1(worst) to 5(best)
  12. Physical health or emotional problems affected social activities,score 1(worst) to 5(best)
Patient involvement | Up to 20 months and two weeks
  Data collected by questionnaire at baseline, 3 and 6 months include:
  Health Education Impact Questionnaire (HEIQ): positive and active engagement in life.
  The heiQ contains 40 items with 4 response categories, scores from 1 (worst) to 4 (best).
Location and setting for physical activity | Up to 44 months and two weeks
  Data collected by a singe item question at baseline,12 and 24 months;
  A multiple choice question with a single answer:
  Are you physically active:
  * on your own?
  * In sports associations?
  * In adult learning school?
  * In other settings?
  Data collected by phone calls 1 and 3 months after end rehabilitation;
  A multiple choice question with a single answer:
  Are you physically active:
  * on your own?
  * In sports associations?
  * In adult learning school?
  * In other settings?

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Birke, Ph.D., Principal Investigator — Center for Clinical Research and Prevention
Locations (1):
- Center for Clinical Research and Prevention, Frederiksberg, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birke H, Foxvig I, Burns K, Toft U, Hansen ABG, Hauge PI, Foghmar S, Mindegaard RB, Jakobsen LM. Heart Rehabilitation for All (HeRTA): Protocol for a feasibility study and pilot randomized trial. PLoS One. 2022 Jun 17;17(6):e0270159. doi: 10.1371/journal.pone.0270159. eCollection 2022. PMID 35714121